CLINICAL TRIAL: NCT01667822
Title: Cognitive Behavioral Therapy, Guided Self Help Versus Individual Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Self help CBT
Record Dates: First submitted 2012-08-10; First posted 2012-08-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Anxiety Disorders; Major Depression; Stress Disorders; Primary Insomnia
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major; Stress Disorders, Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continued guided self help CBT (Active Comparator): Continued guided self help CBT. Participants will receive CBT through self-help books with minimal therapist contact (3 sessions in total).
  Interventions: Behavioral: Continued self help CBT
- CBT individual therapy (Experimental): After the initial face of self help CBT, patients in this arm receive individual CBT. The cognitive behavior therapy used in the study will be based on the protocols with best empirical support.The therapy is delivered by the same psychologist as in the first face and the second face builds on the learning's from the first face.
  Interventions: Behavioral: Individual CBT

INTERVENTIONS:
Behavioral: Continued self help CBT — After the initial Guided self help, patients in this arm continue the same self help program with 1 additional guiding session.
  Arms: Continued guided self help CBT
Behavioral: Individual CBT — After the initial face of self help CBT, patients in this arm receive individual CBT. The cognitive behavior therapy used in the study will be based on the protocols with best empirical support.The therapy is delivered by the same psychologist as in the first face and the second face builds on the learning's from the first face.
  Arms: CBT individual therapy

SUMMARY:
Background: Studies show that about 1 out of 3 patients in Primary Care suffer primarily from mental health disorders, such as anxiety disorders and depression. Cognitive behavior therapy (CBT) has been shown to be an effective treatment of these disorders. Despite the strong evidence for CBT there is a lack of evidence-based psychological treatment in primary care. For various reasons, the progress of research has not affected clinical practice. For successful implementation of CBT in primary care cost-effective therapies, access to therapists with proper training and supervision, evidence-based manuals and management that support the implementation is needed.

Aim: The aim of this trial is to evaluate a stepped care model with CBT in primary care. All patients are first treated with self-help CBT (N = 400). Patients that do not improve after treatment (9 weeks) are randomized to individual CBT or continued self-help treatment. Based on published studies 2/3 is expected to be improved after self-help and therefore do not undergo randomization. 1/3 (n = 133) who didn´t respond to treatment is randomized to individual CBT (N = 67) or continued self-help treatment (N = 67).

ELIGIBILITY:
Inclusion Criteria:

* Have an anxiety disorder diagnosis (obsessive compulsive disorder, social phobia, panic disorder, generalized anxiety disorder), or/and major depression, or/and maladaptive stress reaction, or/and primary insomnia Clinician severity rating scale 2-6

Exclusion Criteria:

* A higher score than 6 on the Clinician severity rating scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population | 9 weeks
  Absolute improvement, i.e., symptom level below pre-established cut-offs at 9 weeks, 20 weeks, 26 week follow-up, and 52 week follow-up compared to baseline.
Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population | 20 weeks
  Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population
Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population | 26 weeks
  Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population
Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population | 52 weeks
  Absolute improvement in disorder specific symptoms defined as closer to healthy than to clinical population or 2 standard deviations from clinical population

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale-Self-report (MADRS-S) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in MADRS-S at post-treatment, 26 week follow-up, and 52 week follow-up
Work ability index (WAI) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in WAI at post-treatment, 26 week follow-up, 52 week follow-up
Insomnia Severity Index (ISI) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in ISI at post-treatment, 26 week follow-up, and 52 week follow-up
Health Anxiety Inventory (HAI) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in HAI at post-treatment, 26 week follow-up, and 52 week follow-up
Perceived Stress Scale (PSS) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in PSS at post-treatment, 26 week follow-up, and 52 week follow-up
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in TIC-P at post-treatment, 26 week follow-up, and 52 week follow-up
Quality of Life Inventory (QOLI) | Baseline, post-treatment (20 weeks), 26 feel follow-up, 52 week follow-up
  Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
EuroQol-5 dimension (EQ5D) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in EQ5D at post-treatment, 26 week follow-up, and 52 week follow-up
Sheehan Disability Scales (SDS) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Baseline, post-treatment (variable depending on disorder), 26 week follow-up, 52 week follow-up
Self-rated health 5 (SRH-5) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in SRH-5 at post-treatment, 26 week follow-up and 52 week follow-up
Obsessive Compulsive Inventory-Revised (OCI-R) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in OCI-R at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Liebowitz Social Anxiety Scale Self-report (LSAS-SR) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in LSAS-SR at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Panic Disorder Severity Scale Self-rated (PDSS-SR) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in PDSS-SR at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Penn-State Worry Questionnaire (PSWQ) | Baseline, post-treatment (20 weeks), 26 week follow-up, 52 week follow-up
  Change in PSWQ at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.

OTHER OUTCOMES:
Inflammatory cytokines | Baseline, post-treatment (20 weeks)
  Change in inflammatory cytokines at post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet and Gustavsberg primary care center, Stockholm, Stockholm County, Sweden